CLINICAL TRIAL: NCT01327014
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel Group Study of Lipid-Lowering Effects of XueZhiKang (XZK) in Patients With Hyperlipidemia
Brief Title: Efficacy and Safety Study of Lipid-Lowering Effects of XueZhiKang (XZK) in Patients With Hyperlipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Peking University WBL Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WPU-201
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; Cholesterol; Lipids; Lipoproteins; XueZhiKang; Botanical
MeSH Terms: conditions — Hyperlipidemias | interventions — xuezhikang

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- 1,200 mg/day of XZK group (Experimental)
  Interventions: Drug: XueZhiKang (XZK), a botanic product with multiple components
- 2,400 mg/day of XZK group (Experimental)
  Interventions: Drug: XueZhiKang (XZK), a botanic product with multiple components

INTERVENTIONS:
Drug: XueZhiKang (XZK), a botanic product with multiple components — 4 capsules of study drug twice a day for 12 weeks.
  Arms: 1,200 mg/day of XZK group; 2,400 mg/day of XZK group
Drug: Placebo — 4 capsules twice a day for 12 weeks.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to demonstrate the efficacy of XueZhiKang to improve plasma lipid profile, as compared to placebo, in outpatients with hyperlipidemia.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, placebo-controlled, parallel group study to be conducted in approximately 120 patients with hyperlipidemia in approximately 10 sites in US and China. Patients who satisfy the entry criteria at screening visit will have a 4-week Therapeutic Lifestyle Changes (TLC) diet control period during which all lipid-lowering medications will be discontinued. After the 4-week diet control period, eligible patients will be randomized to one of three treatment groups. The treatment period will last for 12-weeks. Patients will have blood samples collected at 5 time points (screening, baseline, Week 4, Week 8, and Week 12).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with hyperlipidemia as defined by fasting levels of TC ≥ 240 mg/dl and LDL-C ≥ 160 mg/dl but < 190 mg/dl and TG < 400 mg/dl.
2. Patients with a 10-year coronary heart disease risk Framingham Point Score of < 10%.
3. Male or female patients, of any race, at least 18 years of age.
4. Female patients must be postmenopausal as defined by no menstruation for at least 12 months, or surgically sterilized for at least three months prior to beginning the study, or have a negative pregnancy test and agree to avoid pregnancy during the study and one month after the end of the study by using two reliable methods of contraception.
5. Patients must have been informed of all aspects of the study and signed an informed consent form before any study-related activities.
6. Patients must be willing to follow the TLC diet.
7. BMI < 36 kg/m2.
8. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients with myocardial infarction, stroke, transient ischemic attack, cardiovascular surgery or major operations within 6 months prior to screening visit.
2. Patients with percutaneous coronary intervention within 3 months.
3. Patients who have been taken lipid-lowering medications including statins or XZK during the 4 weeks prior to screening visit.
4. Patients with uncontrolled hypertension at the screening visit. Patients on stable antihypertensive medication may be enrolled provided that the medications and dosage remain stable throughout the study.
5. Patients who are taking anticoagulants except aspirin at < 325 mg/day.
6. Patients with liver dysfunction as indicated by a serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) level of > 1.5-times of upper limit of normal (ULN) range, or clinical symptoms.
7. Patients with elevated creatine phosphokinase level (above Upper Limit of Normal range).
8. Patients with renal dysfunction as indicated by a serum creatinine level above ULN range, or clinical symptoms.
9. Patients with gastric or peptic ulcer within 3 months prior to screening visit.
10. Patients with uncontrolled diabetes mellitus as defined by a HbA1c level of > 7.0%.
11. Patients with medical history of hypothyroidism, pancreatitis, cholestasis, nephrotic syndrome, gall bladder disease, or primary biliary cirrhosis. Patients on thyroid replacement therapy at stable doses may be enrolled if clinically euthyroid.
12. Patients with clinically relevant illness within 4 weeks prior to the screening visit that may interfere with the conduct of this study.
13. Patients with a history of alcohol or narcotic substance abuse within two years prior to screening visit.
14. Patients with hypersensitivity to lipid-lowering agents.
15. Patients who have taken another investigational drug within 4 weeks prior to screening visit.
16. Patients with uncontrolled metabolic or endocrine disease knowing to influence lipid values.
17. Patients who are known to be HIV positive.
18. Patients who have a history or presence of active malignancy (other than non-melanoma skin cancer) or clinically significant psychiatric, neurological, respiratory, hematological, or other conditions that in the opinion of investigators might interfere with or contraindicate participation of the patients in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mean percentage change from baseline at week 12 (or the last assessment) on serum low-density lipoprotein cholesterol (LDL-C) level. | Screening, Baseline, Week 4, Week 6, and Week 12

SECONDARY OUTCOMES:
Mean percentage change from baseline at week 12 (or the last assessment on serum total cholesterol (TC) level. | Screening, Baseline, Week 4, Week 6, and Week 12
Mean percentage change from baseline at week 12 (or the last assessment) on serum high-density lipoprotein cholesterol (HDL-C) level | Screening, Baseline, Week 4, Week 6, and Week 12
Mean percentage change from baseline at week 12 (or the last assessment) on serum triglyceride (TG) level. | Screening, Baseline, Week 4, Week 6, and Week 12
Mean percentage change from baseline at week 12 (or the last assessment) on serum non-HDL cholesterol level. | Screening, Baseline, Week 4, Week 6, and Week 12
Mean percentage change from baseline at week 12 (or the last assessment) on serum apolipoprotein A-I (Apo A-I) and serum apolipoprotein-B (Apo-B) and the Apo-B/Apo A-I ratio. | Screening, Baseline, Week 4, Week 6, and Week 12
Mean percentage change from baseline at week 12 (or the last assessment) on the serum TC/HDL-C ratio. | Screening, Baseline, Week 4, Week 6, and Week 12
Percentage of patients who show a LDL-C level of <130 mg/dl or <100 mg/dl at end of the study. | Screening, Baseline, Week 4, Week 6, and Week 12
Safety will be assessed by the incidence of adverse events (AEs), discontinuation due to the AEs, clinically relevant changes on laboratory test results, vital signs, physical examinations, and 12-lead electrocardiograms (ECG). | Screening, Baseline, Week 4, Week 6, and Week 12; ECG and Physical exam only at Screening and Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: David Capuzzi, Principal Investigator — Cardiovascular Medical Associates
Locations (13):
- United States (8):
  - Robert Karns, MD A Medical Corporation, Beverly Hills, California
  - Jellinger and Lerman, MD, Hollywood, Florida
  - Department of Internal Medicine, University of Kansas Medical Center, Kansas City, Kansas
  - Harold E Bays, MD, Louisville, Kentucky
  - Eli M Roth, MD, Cincinnati, Ohio
  - Cardiovascular Medical Associates, Philadelphia, Pennsylvania
  - Osvaldo Brusco, MD, Corpus Christi, Texas
  - Clinical Trial Network, Houston, Texas
- China (5):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Wuhan Union Hospital, Wuhan, Hubei
  - Second Xiangya Hospital of Central-South Univ, Changsha, Hunan
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality